CLINICAL TRIAL: NCT04515550
Title: Longitudinal Biospecimen Collection for Mitochondrial Metabolomics in Huntington's Disease
Brief Title: Mitochondrial Biomarkers in Huntington's Disease
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Case Western Reserve University (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Steven Gunzler, MD, Assistant Professor, Neurology, University Hospitals Cleveland Medical Center
Other Study IDs: 20181082; 1R21NS107897-01A1 (NIH)
Record Dates: First submitted 2020-07-31; First posted 2020-08-17 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Huntington Disease
Keywords: Huntington disease; Huntington's disease; biomarker
MeSH Terms: conditions — Huntington Disease | interventions — Spinal Puncture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples Without DNA — blood and csf specimens for mitochondrial metabolomics
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Huntington's disease (HD): people with HD
  Interventions: Diagnostic Test: lumbar puncture
- Controls without HD: people without HD
  Interventions: Diagnostic Test: lumbar puncture

INTERVENTIONS:
Diagnostic Test: lumbar puncture — Some participants will have an optional lumbar puncture

SUMMARY:
The objective of this study is to discover a panel of mitochondrial metabolomics biomarkers for Huntington's disease.

DETAILED DESCRIPTION:
This investigator-initiated, single-site longitudinal study seeks to assess the utility of mitochondrial metabolomics -- panels of small molecules that affect mitochondrial function -- to diagnose pre-symptomatic, pre-manifest, and symptomatic Huntington's disease and serve as biomarkers for HD severity and progression. It also seeks to demonstrate that this novel biomarker in the blood has comparable value to the same analysis in spinal fluid. This research study involves 3-4 visits over 18 months. Forty volunteers with HD and 25 volunteers without HD will be included. Volunteers who have HD will have a physical examination and blood draw at each study visit. Some participants will also volunteer for optional lumbar puncture.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 85
* Montreal Cognitive Assessment score >10
* HD subjects had onset of HD symptoms after the age of 20
* HD subjects with Diagnostic Confidence Level (DCL) of 0-3 (pre-symptomatic or pre-manifest) must have at least 40 CAG repeats on one HTT allele
* HD subjects with Diagnostic Confidence Level (DCL) of 4 (manifest) must have at least 36 CAG repeats on one HTT allele
* Controls are asymptomatic without family history of HD or have <36 CAG repeats on both HTT alleles with family history of HD

Exclusion Criteria:

* HD subjects who did not already have genetic testing are excluded from this study
* Pregnancy or plans to become pregnant during the study
* Investigational drugs within 3 months of screening visit
* Alcohol or illicit drug abuse or dependence
* Other genetic or neurological disorders
* Other medical or psychiatric illness that in the investigator's judgement will prevent ability to tolerate or undergo study procedures
* For those volunteering for lumbar puncture (LP), bleeding disorders or excessive bleeding, anticoagulation, aspirin if unable to safely stop taking it at least 7 days prior to LP, other antiplatelet medications, inability to tolerate LP, allergy to local anesthetic or chlorhexidine, major lumbar spine deformity, low platelets or abnormal coagulation factors PT/APTT

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of people with HD and controls without HD
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Change in Unified Huntington Disease Rating Scale (UHDRS) and UHDRS sub-sections | At baseline, 9 months, and 18 months
  This is a questionnaire and neurological examination. Lower values are better than higher values.

SECONDARY OUTCOMES:
Change in Montreal Cognitive Assessment (MoCA) | At baseline, 9 months, and 18 months
  Zero to 30 point cognitive scale. Higher values are better than lower values.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Qi, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No